CLINICAL TRIAL: NCT00019513
Title: A Phase I Study of Weekly Gemcitabine in Combination With Infusional 5-Fluorouracil and Oral Calcium Leucovorin in Adult Cancer Patients
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent, Refractory, or Metastatic Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 980143; 98-C-0143; CDR0000066587; NCT00001706 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer; Lung Cancer; Lymphoma; Pancreatic Cancer; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent adult primary liver cancer; advanced adult primary liver cancer; adult primary cholangiocellular carcinoma; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent pancreatic cancer; stage IV esophageal cancer; recurrent esophageal cancer; recurrent colon cancer; stage IV colon cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; cholangiocarcinoma of the gallbladder; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; cholangiocarcinoma of the extrahepatic bile duct; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Lung Neoplasms; Lymphoma; Pancreatic Neoplasms; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Colonic Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Fluorouracil; Gemcitabine; Leucovorin

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining gemcitabine, fluorouracil, and leucovorin in treating patients with recurrent, refractory, or metastatic solid tumors or lymphomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical toxic effects associated with administering sequential gemcitabine followed by fluorouracil with leucovorin calcium in patients with refractory or recurrent or metastatic solid tumors or lymphomas.
* Determine achieved steady-state plasma levels of gemcitabine and fluorouracil in these patients.
* Determine any antitumor activity of this regimen in these patients.
* Determine the pharmacodynamics of gemcitabine and fluorouracil in these patients.

OUTLINE: This is a dose-escalation study of fluorouracil and gemcitabine.

During the first course, patients receive gemcitabine IV over 30 minutes once weekly for 2 weeks followed by one week of rest. During subsequent courses, patients receive gemcitabine as above followed immediately by fluorouracil IV over 24 hours once weekly for 2 weeks. Patients also receive leucovorin calcium orally on days 1 and 8 and IV on days 2 and 9. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Sequential dose escalation of fluorouracil is followed by sequential dose escalation of gemcitabine. Cohorts of 3-6 patients receive escalating doses of fluorouracil and then gemcitabine until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 108 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer that has failed standard therapy or for which no such therapy exists, including, but not limited to:

  * Unresectable primary or recurrent solid tumors (e.g., colon, pancreatic, lung, esophageal, or cholangiocarcinoma)
  * Metastatic disease
  * Lymphoma with no prior high-dose chemotherapy requiring autologous or allogeneic stem cell rescue
* No leukemias
* No CNS metastases or primary CNS malignancies
* No failure on prior gemcitabine therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Transaminases less than 6 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious concurrent medical illness that would preclude study
* No active infections requiring IV antibiotics
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* More than 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (at least 6 weeks for mitomycin or nitrosoureas) and recovered
* At least 3 months since prior suramin
* At least 5 weeks since prior eniluracil (8 weeks prior to start of fluorouracil) and recovered

Endocrine therapy:

* No steroid therapy if utilized for chronic lymphoma therapy
* At least 4 weeks since prior steroidal therapy as disease treatment

Radiotherapy:

* At least 2 weeks since prior radiotherapy to no more than 20% of bone marrow
* At least 4 weeks since prior radiotherapy to 21% or more of bone marrow
* Recovered from prior radiotherapy

Surgery:

* Recovered from prior surgery

Other:

* No concurrent cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 1998-08; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szabo, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wright MA, Schuler B, Szabo E, Grem JL. Sustained partial response of an intra-abdominal desmoid tumor treated with gemcitabine, 5-fluorouracil and leucovorin. Ann Oncol. 2003 Apr;14(4):659-60. doi: 10.1093/annonc/mdg155. No abstract available. PMID 12649120